CLINICAL TRIAL: NCT03633981
Title: Multimodal Assessment of the Neurological Prognosis of Patients With Brain Lesions on ExtraCorporeal Life Support
Acronym: NeuroECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ELLOUZE 2018 Neuro ECMO
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-08

CONDITIONS: Brain-injured Patients on Extracorporeal Life Support
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical examinations — Collection of data from the following tests at H0 (as soon as the ECLS is put in place), H12 (within 12 hours following stabilisation of the dynamic state), H24 and every day until complete neurological recovery:
  * right and left pupillometry (3 times)
  * BIS values
  * right and left NIRS values
  * right and left transcranial Doppler
  * neurological clinical examination
Other: neurological assessment when a neurological event occurs — next neurological event:
  * seizures
  * pupillary asymmetry
  * myoclonias
  * brain stem reflex abnormalities
  * osteotendinous reflex abnormalities
Other: mortality assessment — to 28 days

SUMMARY:
It seems of the greatest importance to evaluate the neurological prognosis of patients with brain lesions after cardiorespiratory arrest or circulatory failure requiring circulatory assistance.

However, to date, there is no clinical or paraclinical diagnostic test to reliably assess the future of these patients.

The objective of this study is to highlight the clinical and imaging factors for establishing a neurological prognosis in patients at risk of brain lesions under ExtraCorporeal Life Support (ECLS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain lesions on veno-arterial circulatory support after cardiac arrest or cardiogenic shock who require at least 24 hours of sedation

Exclusion Criteria:

* Extubation expected within the first 24 hours of management
* Minor patient
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain lesions on veno-arterial ECLS after cardiac arrest or cardiogenic shock, requiring at least 24 hours sedation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Early mortality assessment | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Omar ELLOUZE, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (1):
- Chu Dijon Bourogne, Dijon, France